CLINICAL TRIAL: NCT05108675
Title: Elucidating the Dynamics and Impact of the Gut Microbiome on Maternal Nutritional Status During Pregnancy
Brief Title: Microbiome and Malnutrition in Pregnancy (MMiP)
Acronym: MMiP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); University of Toronto (Other); University of Calgary (Other); Dalhousie University (Other); University of Alberta (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor Zulfiqar A Bhutta MBBS, FRCPCH, FAAP, PhD, Aga Khan University
Other Study IDs: 51950
Record Dates: First submitted 2021-09-22; First posted 2021-11-05 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-07

CONDITIONS: Weight Gain, Pregnancy; Microbial Colonization; Pregnancy Related; Pregnancy Loss; Pregnancy Complications; Pregnancy; Parasitic Disease; Parasitic Disease; Microbial Disease; Infant Malnutrition; Malnutrition; Malnutrition in Pregnancy; Breastfeeding
Keywords: Maternal Malnutrition, Gut Dysbiosis, Infant Health
MeSH Terms: conditions — Gestational Weight Gain; Communicable Diseases; Pregnancy Complications; Parasitic Diseases; Infant Nutrition Disorders; Malnutrition; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood samples will be collected from mother and infant.
  Participants will have the option to have their blood samples biobanked for future genetic testing (This would be a separate study application in the future).
  More information on sample analysis can be found in section 10 of the protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nutritional status during pregnancy plays an important role in maternal health and birth outcomes. While few factors impacting nutritional status during pregnancy have been identified, studies of undernutrition in children have revealed a key role for the gut microbiome. Remarkably, studies examining the dynamics of the maternal gut microbiome before and during pregnancy and its impact on birth outcomes are limited.

This study is being conducted to investigate how a mother's nutritional status and her gut microbiome during pregnancy contribute to the birth outcomes and health of her baby. The gut microbiome is the totality of microorganisms (e.g. bacteria, viruses, fungi) living in the gastrointestinal tract. This study will focus on married pregnant women 24 years and younger living in Matiari District in Pakistan. The focus is on younger women due to their vulnerability to undernutrition. Pregnant participants, and upon delivery, their newborns will be followed throughout pregnancy and for a year afterwards. Throughout this period, the investigators will collect stool samples, rectal swabs, blood samples, health assessments, nutritional and dietary assessments and birth/ labour details. The goal is to define the relationship between a mother's nutritional status and her microbiome dynamics during pregnancy and how they contribute to the birth outcomes and growth of her newborn. Investigators hypothesizes that alterations of the microbiota in the maternal gut (dysbiosis) is exacerbated by nutritional status or pathogen exposure during pregnancy. This impacts weight gain because of impaired nutrient absorption, and can lead to corresponding negative birth outcomes.

DETAILED DESCRIPTION:
This project represents the first systematic investigation of the impact of the microbiome on nutritional status during pregnancy in young women and directly aligns with global health initiatives focused on this vulnerable cohort. The goal of the study is to define the relationships between host nutritional status and microbiome dynamics during pregnancy and how they contribute to birth outcomes. The gut microbiome has a profound influence on host nutritional status. Dysbiosis (loss of diversity/beneficial microbes and gain of pathobionts) has emerged as a major factor in the development of undernutrition. Despite the importance of nutrition during pregnancy, few studies have examined the role of the microbiome on maternal health and birth outcomes. Further, little is known concerning the influence of enteric eukaryotic microbes, such as parasites, on the bacterial microbiome and host nutrition.

At the core of this study are two complementary cohorts of young women that provide an exceptional opportunity to obtain longitudinal samples to monitor the dynamic relationships between microbiome community structure and function with gut health and host nutritional status. This registration is for the Matiari, Pakistan cohort of the study, where there is known to be a high prevalence of undernutrition among young women. This cohort is expected to yield insights into the influence of eukaryotic microbes that are often viewed as asymptomatic. The target demographic of the study is young, married mothers, ≤24 years in Matiari District within the province of Sindh, Pakistan. Matiari District is representative of rural settings in Pakistan The investigators have identified this younger demographic due to the lack of knowledge on the microbiome of young women, and their vulnerability to undernutrition. A second complementary cohort will be based Toronto, Canada. This project will yield insights into the relationships between prokaryotic and eukaryotic microbes in the gut and their associations with maternal health and birth outcomes.

The central hypothesis of the study is that alterations of the microbiota in the maternal gut (dysbiosis) exacerbated by nutritional status or pathogen exposure during pregnancy, impacts weight gain because of impaired nutrient absorption, leading to corresponding negative birth outcomes.

The study will be a prospective, longitudinal, observational study to investigate the impact and relationship between prokaryotic and eukaryotic microbes in the gut and their association with maternal health and birth outcomes among married young women ≤24 years residing in Matiari District. . The study will aim to recruit 400 women into two groups based on BMI at time of recruitment (normal BMI will be defined as between 20 and 24.9 kg/m2 and low BMI will be defined as less than 20 kg/m2). With a goal of having 200 participants within the normal BMI group and 200 participants within the low BMI group. Although this is the recruitment aim, in the event that the investigators are unable to recruit 200 women with a low BMI, more women will be recruited that fall within the normal BMI range. The study will follow women and their infants over the course of their pregnancy and for a year postpartum, collecting stool, rectal and blood samples, nutritional information, heath assessments, anthropometric measurements and empowerment metrics at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided
* Married female aged 17-24 years
* In good general health, with no comorbidities
* Absence of COVID19 symptoms
* Intend to comply with study procedures and follow up

Exclusion Criteria:

* Women who do not meet the enrollment age criteria
* Women participating in interventional clinical trials
* Women who intend to leave the study area
* Women who cannot comply with study procedure's and follow-up
* Illness and other co-morbidities
* Signs of potential COVID19 infection
* BMI higher than 24.9 kg/m2
* Women who already have a member of their household participating
* Women who have taken antibiotics within the past 3 months
* Women who are past 16 weeks post- conception

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Biological sex: as the study's primary aim is to investigate pregnancy, participation will be restricted to participants who are biologically female. However, the study is inclusive with respect to gender, including both cis-gendered and trans-gendered participants (biological female-to-male).
Study Population: This study will examine young, married women ≤24 years living in Matiari District, Pakistan. The investigators focus on younger women, due to the lack of knowledge about their microbiome and their vulnerability to undernutrition
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess if alterations of the microbiota in the maternal gut (dysbiosis) are corelated with changes in maternal gestational weight gain | 8-20 weeks post-conception, 30-34 weeks post-conception
  The primary endpoint will be the change in maternal gestational weight gain (GWG) during pregnancy, measured between the first (8-16 weeks post-conception) and second time point (30-34 weeks post-conception)
To determine the correlation between maternal microbiome dysbiosis during pregnancy and birth weight. | At birth
  The primary endpoint will be change in birthweight measured in kilograms.
To determine the correlation between maternal microbiome dysbiosis during pregnancy and infant growth | 3month, 6month and 12month postpartum
  The primary endpoint will be change in WHO z-scores during first year of infant's life. These z-scores will be calculated for weight (measured in kg), length and head circumference (measured in cm).

SECONDARY OUTCOMES:
Anthropometrics | 8-16 weeks post-conception, 30-34 weeks post-conception, delivery, 3-months post-partum, 6 months post-partum and 12 months post-partum ]
  Maternal BMI
Anthropometrics: Maternal middle upper arm circumference | 8-16 weeks post-conception, 30-34 weeks post-conception, 3-months post-partum,and 12 months post-partum
  Measured in cm
Anthropometrics: Maternal triceps skinfold thickness | 8-16 weeks post-conception, 30-34 weeks post-conception, 3-months post-partum, and 12 months post-partum
  Measured in mm
Anthropometrics: Maternal height | 8-16 weeks post conception, 30-34 weeks post conception, delivery, 3 months post-partum and 12 months post partum
  measured in cm
Anthropometrics: Maternal weight | 8-16weeks post conception, 30-34 weeks post conception, delivery, 3 months post-partum and 12 months post-partum
  measured in kg
Maternal blood biomarker-1 | 8-16 weeks post-conception, 30-34 weeks post-conception, and 12 months post-partum
  Concentration of HB in g/dL, marker of anemia.
Maternal blood biomarker-2 | 8-16 weeks post-conception, 30-34 weeks post-conception, and 12 months post-partum
  Level of MCV in whole blood measured in femtoliters (fL).
Maternal blood biomarker-3 | 8-16 weeks post-conception, 30-34 weeks post-conception, and 12 months post-partum
  Concentration of Ferritin in serum measured in ng/mL, marker of iron stores in blood.
Maternal blood biomarker-4 | 8-16 weeks post-conception, 30-34 weeks post-conception, and 12 months post-partum
  Concentration of CRP in blood, measured in mg/dL, marker of inflammation .
Infant blood biomarker-1 | 1 year infant age
  Concentration of HB in g/dL, marker of anemia.
Infant blood biomarker-2 | 1 year infant age
  Level of MCV in whole blood measured in femtoliters (fL).
Infant blood biomarker-3 | 1 year infant age
  Concentration of Ferritin in serum measured in ng/mL, marker of iron stores in blood.
Infant blood biomarker-4 | 1 year infant age
  Concentration of CRP in blood, measured in mg/dL, marker of inflammation .
Infant sex | At birth
  Male Female
Infant morbidity | at 3 months, 6 months and 12 months
  Assessed through infant health assessment questionnaire
Maternal morbidity | 8-16 weeks post-conception, 30-34 weeks post-conception, 3 months post-partum, 6 months post-partum and 12 months post-partum
  Assessed through health assessment questionnaire
Infant growth: weight | within 72 hours of birth, 3 months, 6 months and 12 months
  Measured in kg
Infant growth: length | within 24 hours of birth, 3 months, 6 months and 12 months
  Measured in cm
Infant growth: head circumference | within 72 hours of birth, 3 months, 6 months and 12 months
  Measured in cm
Infant growth: mid upper arm circumference | within 72 hours of birth, 3 months, 6 months and 12 months
  Measured in cm
Infant growth: triceps skinfold thickness | within 72 hours of birth, 3 months, 6 months and 12 months
  Measured in mm
Gestational age at birth | Within 72 hours of birth
  Measured in weeks
Maternal age | 8-16 weeks post conception
  Age between 17-24 years documented through national ID card, school certificate or through maternal recall
Breast feeding | at birth within 72 hours, 3 months, 6 months and 12 months
  amount and initiation of breast feeding, top milk, formula milk and complementary feeding Based off of WHO 2010 Guidelines: Indicators for assessing infant and young child feeding practices (Part 2 Measurement)
Reported Maternal medicinal use | 8-16 weeks post-conception, 30-34 weeks post-conception, 3-months post-partum, 6 months post-partum and 12 months post-partum
  Questionnaire
Reported Infant medication use | at birth within 72 hours, 3 months, 6 months and 12 months
  Questionnaire
Maternal dietary intake Assessed through ASA 24 HR Dietary Recall system, completed 2x each time point | Baseline 8-16 weeks post conception, 30-34 weeks post conception and 12 months post partum
  Assessed through ASA 24 HR Dietary Recall system
Dietary diversity | Baseline 8-16 weeks post conception, 30-34 weeks post conception, 3 months post-partum and 12 months post partum
  Minimum Dietary Diversity Score for Women (MDD-W)
Household annual food insecurity | 3 months post-partum and 12 months post-partum
  Food insecurity will be assessed using the Household Food Insecurity Access Scale (HFIAS)
Generalized Self-efficacy | 3 months post-partum and 12 months post partum
  Self-efficacy will be measured using the Generalized Self-Efficacy scale, developed by Schwarzer and Jerusalem. A 10 item psychometric scale.
Perceived decision making | 3 months post-partum and 12 months post partum
  Questions pertaining to perceived decision-making are from the Pakistan Demographic and Health Survey (PDHS)
Perceived social support | 3 months post-partum and 12 months post partum
  Perceived social support will be measured using the Multi-dimensional Scale of Perceived Social Support (MSPSS), developed by Zimet et al.
Maternal demographics | Baseline 8-16 weeks post-conception
  Questions pertaining to demographic data are adapted from the Pakistan Demographic and Health Survey (PDHS)
Food insecurity | Baseline 8-16 weeks post conception, 3 months post partum and 12 months post partum
  Questionnaire developed by Hager, E.R., et al., Development and validity of a 2-item screen to identify families at risk for food insecurity.
Perceived parental stress | 3 months post-partum and 12 months post partum
  Perceived parental stress will be measured using the Perceived Stress Scale (PSS-10)
Preterm Births | At birth within 72 hours
  Gestational age at birth in weeks
Small for gestational age | At birth within 72 hours
  Small-for-gestational-age (<10th percentile of weight-for-gestational-age and sex as defined by Intergrowth standards)
Large for gestational age | At birth within 72 hours
  >90th percentile of weight-for-gestational-age and sex as defined by Intergrowth standards)
Delivery Assessment | at birth within 72 hours of birth
  Questionnaire, mode of delivery, place of birth and other description around delivery
Infant dietary intake | Infant age 1 year
  NutricheQ Questionnaire: a tool designed for toddlers aged 1 to 3 years of age, with a focus on markers for inadequate or excessive intake and dietary imbalances
Maternal stool biomarkers-1 | At baseline 8-16 weeks post conception and 30-34 weeks post conception
  Level of Calprotectin in stool a marker of intestinal inflammation, measured in μg/g.
Maternal stool biomarkers-2 | At baseline 8-16 weeks post conception, 30-34 weeks post conception
  Concentration of Claudin 15 in stool a marker of intestinal permeability measured in ng/mL.
Maternal stool biomarkers-3 | At baseline 8-16 weeks post conception and 30-34 weeks post conception
  Concentration of Lipocalin in stool, a marker of gut inflammation, measured in μg/mL.
Maternal: incidence of pathobionts | Baseline, 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  As identified through 16S, 18S and ITS rDNA surveys
Infant: incidence of pathobionts | 3 and 12 month
  As identified through 16S, 18S and ITS rDNA surveys
Maternal: metabolomic profile of stool [Metabolites involved in central metabolism as analysed by Mass Specttrometry] | Baseline, 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  Analysis of the core metabolites involved in central metabolism. These metabolites will be analysed through Mass Spec and include short chain fatty acids, amino acids, intermediates in energy metabolism and nucleotide biosynthesis
Maternal gut bacteria profile | Baseline, 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  Measured through 16S rDNA sequence surveys
Maternal: blood metallomics profile | Baseline, 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  Measured through ICP-MS (https://www.metabolomicscentre.ca/new_service/25) - TMIC platform of metabolmics
Infant: blood metallomics profile | Infant age 1 year
  as measured through ICP-MS (https://www.metabolomicscentre.ca/new_service/25) Through TMIC platform
Infant: gut bacterial profile | 3 month and 12 month
  Measured through 16S rDNA sequence surveys
Maternal metabolic pathway expression profile | Baseline 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum
  as measured through whole microbiome RNASeq (metatranscriptomics)
Infant eukaryotic microbiome profile | 3 & 12 Months
  as measured through 18S and ITS rDNA sequence surveys
Maternal eukaryotic microbiome profile | Baseline 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum ]
  as measured through 18S and ITS rDNA sequence surveys
Maternal bacterial gene expression profile | Baseline 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum ]
  as measured through whole microbiome RNASeq (metatranscriptomics) - The output of these analyses are readouts of microbial gene expression detailing biochemical activities as well as the taxa responsible.
Maternal: microbiome taxonomic alpha and beta diversity | Baseline 8-16 weeks post conception, 30-34 weeks post conception, 3 months post partum and 12 months post partum ]
  To define taxonomic diversity, species profiles from 16S, 18S and ITS rDNA data will be clustered to identify differences in community structure across samples. Alpha diversity will be measured through indices such as Chao, Shannon and Simpson indices. Beta diversity will be measured through standard indices such as Bray-Curtis distances.
Infant: microbiome taxonomic alpha and beta diversity | 3 and 12 months postpartum
  To define taxonomic diversity, species profiles from 16S, 18S and ITS rDNA data will be clustered to identify differences in community structure across samples. Alpha diversity will be measured through indices such as Chao, Shannon and Simpson indices. Beta diversity will be measured through standard indices such as Bray-Curtis distances.

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar Bhutta, Principal Investigator — Aga Khan University
Locations (1):
- Research and Training Centre Matiari, Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
In addition to publishing findings in open access journals, the investigators will ensure all sequences and metabolomics datasets are deposited in appropriate public repositories of those who consented for this deidentified data sharing. SOPs, pathogen samples and statistical methods developed through this project will be shared with the IMPACTT research core (https://www.impactt-microbiome.ca/). Microbiome sequence data will be uploaded on the National Centre for Biotechnology Information (NCBI).
  The NCBI acts as a central data repository for sequence data. In line with publication standards, the investigators are required to provide access to users who may wish to follow up on analyzing the microbiome data for their own purposes.
  The sample analysis information, including the sequencing data and metabolomics data will be de-identified and the patient sequence data will be removed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All sequence and metabolomics data will be made available within 12 months of study completion Supporting information will be shared at time of request
Access Criteria: Supporting information will be shared upon request Sequence and metabolomics datasets will be made available without restriction

REFERENCES:
- [Derived] Wasan Y, Baxter JB, Spiegel-Feld C, Begum K, Rizvi A, Iqbal J, Hulst J, Bandsma R, Suleman S, Soofi S, Parkinson J, Bhutta ZA. Elucidating the dynamics and impact of the gut microbiome on maternal nutritional status during pregnancy, effect on pregnancy outcomes and infant health in rural Pakistan: study protocol for a prospective, longitudinal observational study. BMJ Open. 2024 Aug 12;14(8):e081629. doi: 10.1136/bmjopen-2023-081629. PMID 39134435

DOCUMENTS (2):
  • Study Protocol (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT05108675/Prot_000.pdf
  • Informed Consent Form (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT05108675/ICF_001.pdf